CLINICAL TRIAL: NCT06962787
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1 in Combination With Tyrosine Kinase Inhibitor (TKI) With or Without Pembrolizumab (BL-B01D1+TKI±Pembrolizumab) in Patients With Locally Advanced or Metastatic Renal Cancer
Brief Title: A Study of BL-B01D1+TKI±Pembrolizumab in Patients With Locally Advanced or Metastatic Renal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-204-13
Record Dates: First submitted 2025-04-28; First posted 2025-05-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Axitinib; lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1+TKI±Pembrolizumab (Experimental): Participants receive BL-B01D1+TKI±Pembrolizumab in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: Axitinib; Drug: Lenvatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: Axitinib — Oral administration, and twice daily with an interval of 12 hours.
Drug: Lenvatinib — Oral administration, and once daily.
Drug: Pembrolizumab — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This Phase II study is a clinical study to explore the efficacy and safety of BL-B01D1 in combination with tyrosine kinase inhibitor (TKI) with or without pembrolizumab (BL-B01D1+TKI±Pembrolizumab) in patients with locally advanced or metastatic renal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject volunteered to participate in the study and signed an informed consent;
2. Male or female aged ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. ECOG score 0 or 1;
5. Patients with locally advanced or metastatic renal cell carcinoma confirmed by histopathology and/or cytology;
6. Agree to provide archived tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. Organ function level must meet the requirements;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. Fertile female subjects, or male subjects with fertile partners, must use highly effective contraception from 7 days before the first dose until 7 months after the first dose. Female subjects of childbearing potential had to have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Chemotherapy, biological therapy and other anti-tumor therapies have been used within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral drugs such as fluorouracil;
2. Prior treatment with an ADC drug containing a camptothecin derivative (topoisomerase I inhibitor) as a toxin;
3. Use of immunomodulatory drugs within 14 days before the first dose of study drug;
4. The history of severe cardiovascular and cerebrovascular diseases within six months before screening;
5. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
6. Active autoimmune and inflammatory diseases;
7. Systemic corticosteroids or immunosuppressive agents are required within 2 weeks before the first dose;
8. Other malignant tumors within 5 years before the first dose;
9. A history of non-infectious ILD requiring steroid treatment, or current ILD/interstitial pneumonia or suspected ILD;
10. Poorly controlled diabetes before starting study treatment; Severe complications of diabetes mellitus;
11. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
12. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
13. Patients with active central nervous system metastasis;
14. Patients with massive or symptomatic effusions or poorly controlled effusions;
15. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to BL-B01D1 or any excipients of pembrolizumab;
16. Previous history of allogeneic stem cell, bone marrow or organ transplantation;
17. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
18. Had a serious infection within 4 weeks before the first dose of study drug; There was pulmonary infection or active pulmonary inflammation at the time of screening;
19. Had participated in another clinical trial within 4 weeks before the first dose (calculated from the time of the last dose);
20. With a history of psychotropic drug abuse and inability to quit or a history of severe neurological or psychiatric illness;
21. Imaging examination showed that the tumor had invaded or wrapped the large thoracic vessels;
22. Serious unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
23. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
24. Subjects scheduled to receive live vaccine or within 28 days before the first dose;
25. Patients with other serious physical and laboratory abnormalities or poor compliance that may increase the risk of participating in the study, or interfere with the results of the study, and patients who were deemed by the investigators to be unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.
Frequency of Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  Frequency of TEAE will be investigated. TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BICR is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China